CLINICAL TRIAL: NCT07242066
Title: Effects of Dietary Nitrate and Vitamin C Co-supplementation on Blood Pressure and Endothelial Function in Overweight Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Kostas Tsintzas, Professor of Human Physiology, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FHMS 128-0224
Record Dates: First submitted 2024-12-05; First posted 2025-11-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Blood Pressure
Keywords: Cardiovascular disease; endothelial function; nitrate; Vitamin C
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo beetroot juice and tablet
  Interventions: Dietary Supplement: Nitrate-depleted beetroot juice plus placebo tablet
- Beetroot juice + Vitamin C (Experimental): Beetroot juice and Vitamin C
  Interventions: Dietary Supplement: Beetroot juice plus vitamin C tablet
- Beetroot juice + placebo (Experimental): Beetroot juice + placebo tablet
  Interventions: Dietary Supplement: Beetroot juice plus placebo tablet

INTERVENTIONS:
Dietary Supplement: Beetroot juice plus vitamin C tablet — Concentrated beetroot juice (70 ml in the morning before breakfast and 70 ml in the evening before dinner) plus Vitamin C tablets (500mg/tablet)
  Arms: Beetroot juice + Vitamin C
Dietary Supplement: Beetroot juice plus placebo tablet — Concentrated beetroot juice (70ml in the morning and 70 ml in the evening) plus placebo tablets (containing 500 mg of the non-nutritive sweetener aspartame)
  Arms: Beetroot juice + placebo
Dietary Supplement: Nitrate-depleted beetroot juice plus placebo tablet — nitrate-depleted beetroot juice (70ml in the morning and 70 ml in the evening) plus placebo tablets (containing 500 mg of the non-nutritive sweetener aspartame)
  Arms: Placebo

SUMMARY:
The investigators have shown in two short-term studies in healthy, young participants that the combined supplementation of inorganic nitrate with vitamin C has beneficial effects on blood pressure and blood vessel wall stiffness. However, the effects of the combined supplementation have not been tested in individuals at greater cardiovascular disease risk. The investigators would like to show whether inorganic nitrate and vitamin C will produce greater effects on blood pressure and endothelial function when compared to inorganic nitrate alone versus the placebo treatment in people at greater risk of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Participant is willing and able to comply with the requirements of the study protocol.
* Non-smoking men and women.
* Aged between 50-75 years.
* Overweight and obese (BMI: over 25.0 kg/m2).

Exclusion Criteria:

* Having taken part in a research study in the last 3 months involving invasive procedures or an inconvenience allowance.
* Vegetarian.
* Smoking.
* Resting systolic blood pressure greater than 160 mmHg; diastolic blood pressure greater than 100 mmHg.
* Active cancer and any diagnosis of malignant cancer in the last 5 years.
* Excessive alcohol intake (>21 units per week).
* Allergy or intolerance to the intervention food (Beetroot juice).
* Diagnosis of chronic or acute metabolic and inflammatory conditions that may interfere with the study outcomes.
* Major surgical operations.
* Use of prescribed psychiatric drugs (antidepressants, sedatives, antipsychotics), diuretics, organic nitrates, statins and proton pump inhibitors.
* Use of prescribed hormonal therapies (oestrogens, thyroxin, and progesterone), anti-hypertensive (Calcium++ channel blockers, beta-blockers, and angiotensin-converting-enzyme (ACE) inhibitors), only if the prescription had started, or the dose had been started/changed, in the previous three months.
* Non-prescribed dietary supplements if not stopped at least for 2 weeks before starting the trial.
* Use of the mouthwash during the study was not allowed as it interferes with the conversion of oral nitrate into nitrite.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Pre, 24 hours, 48 hours and 72 hours after supplementation
  Resting diastolic and systolic blood pressure using portable automated monitor
Cardiac function | Pre and post 3 days of supplementation
  Resting cardiac function using a non-invasive methodology (Finometer)

SECONDARY OUTCOMES:
Flow-mediated dilation | Pre and post 3 days of supplementation
  Assess endothelial function through changes in brachial artery diameter in response to reactive hyperaemia using high-resolution B-mode ultrasound.
Saliva nitrate concentration | Pre and post 3 days supplementation
  Colorimetric assays based on the Griess reaction will be used to measure nitrate concentration in saliva samples
Urinary nitrate concentration | Pre and post 3 days supplementation
  Colorimetric assays based on the Griess reaction will be used to measure nitrate concentration in urine samples
Saliva nitrite concentration | Pre and post 3 days supplementation
  Colorimetric assays based on the Griess reaction will be used to measure nitrite concentration in saliva samples
Urine vitamin C concentration | Pre and post 3 days supplementation
  A colorimetric assay kit will be used to measure vitamin C in urine samples
Urine 8-isoprastane concentration | Pre and post 3 days supplementation
  An Enzyme Linked Immuosorbant assay will be used to determine 8-isoprostane concentrations in urine.

CONTACTS AND LOCATIONS:
Locations (1):
- David Greenfield Human Physiology Lab, Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deanfield JE, Halcox JP, Rabelink TJ. Endothelial function and dysfunction: testing and clinical relevance. Circulation. 2007 Mar 13;115(10):1285-95. doi: 10.1161/CIRCULATIONAHA.106.652859. No abstract available. PMID 17353456
- [Background] Forstermann U. Nitric oxide and oxidative stress in vascular disease. Pflugers Arch. 2010 May;459(6):923-39. doi: 10.1007/s00424-010-0808-2. Epub 2010 Mar 21. PMID 20306272
- [Background] Gori T, Munzel T. Oxidative stress and endothelial dysfunction: therapeutic implications. Ann Med. 2011 Jun;43(4):259-72. doi: 10.3109/07853890.2010.543920. Epub 2011 Feb 1. PMID 21284528